CLINICAL TRIAL: NCT02943369
Title: Cangrelor Administration Following Ticagrelor Loading vs Ticagrelor Loading Alone in ST Segment Elevation Myocardial Infarction Patients: A Randomized, Pharmacodynamic Study
Brief Title: Cangrelor Following Ticagrelor Loading vs Ticagrelor Loading Alone in STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Attikon Hospital (Other)
Collaborators: AHEPA University Hospital (Other); University Hospital, Alexandroupolis (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, National and Capodestrian University of Athens, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS13616
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: STEMI
Keywords: cangrelor; ticagrelor; P2Y12 receptor antagonist; acute myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Ticagrelor; cangrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor (Experimental): Ticagrelor will be followed by Cangrelor
  Interventions: Drug: Ticagrelor 180 mg loading dose; Drug: Cangrelor 30 mcg/kg bolus + 4 mcg/kg/min
- Ticagrelor (Active Comparator): Ticagrelor only
  Interventions: Drug: Ticagrelor 180 mg loading dose

INTERVENTIONS:
Drug: Ticagrelor 180 mg loading dose — Ticagrelor 180 mg
  Other Names: Ticagrelor 180 mg
Drug: Cangrelor 30 mcg/kg bolus + 4 mcg/kg/min — Intravenous Cangrelor 30 mcg/kg bolus + 4 mcg/kg/min for 2 hours
  Other Names: Cangrelor bolus and infusion
  Arms: Cangrelor

SUMMARY:
Platelets and thrombus formation play a key role in the pathogenesis of acute coronary artery occlusion and subsequent myocardial infarction. Apart from mechanically opening the occluded artery with angioplasty, adjunctive antiplatelet treatment is of utmost importance. However, orally administered antiplatelet agents exhibit a delay in their onset of action in the setting of acute myocardial infarction and angioplasty is mostly performed without adequate platelet inhibition. Cangrelor is an intravenous antiplatelet agent which can provide almost immediate strong platelet inhibition. The investigators aim to compare a strategy of cangrelor administered on top of ticagrelor-an oral antiplatelet agent- vs ticagrelor alone, on their efficacy to inhibit platelet function in the early hours of an acute myocardial infarction.

DETAILED DESCRIPTION:
A rapid and consistent platelet inhibition represents the cornerstone of pharmacological treatment in the early hours of ST-segment elevation myocardial infarction (STEMI) with expected improvement in outcome. Current practice guidelines recommend administration of a loading dose (LD) of an oral P2Y12 receptor antagonist as early as possible or at the time of percutaneous coronary intervention (PCI) or at first medical contact.

Pharmacodynamic data have clearly shown a delay in the onset of action when prasugrel or ticagrelor are administered in patients with STEMI - compared to what is obtained in stable or acute coronary syndrome (ACS) patients-, which is most likely caused by an impaired absorption. Peri-interventional platelet inhibition is therefore suboptimal in most cases of timely performed primary PCI, even when novel oral antiplatelet agents with faster than clopidogrel action are used. Modifications of the loading dose or antiplatelet pre-hospital administration may only partially 'bridge the gap" in platelet inhibition.

On the other hand, cangrelor is a parenteral P2Y12 antagonist, with a rapid -within minutes- onset of action, able to provide very strong and consistent platelet inhibition and with rapid offset of action- within 60 min of infusion discontinuation. In the CHAMPION PHOENIX (Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition) trial cangrelor reduced the incidence of ischemic events, without increasing the incidence of severe bleeding. Ticagrelor is an oral antiplatelet agent which has been reported that can be given before or during infusion of cangrelor without attenuation of cangrelor's pharmacodynamic effects, while the pharmacodynamic effects of ticagrelor are preserved when ticagrelor is given during infusion of cangrelor. It seems therefore, that ticagrelor has favorable characteristics for patients intended to receive cangrelor.

In the present study, in STEMI patients undergoing primary PCI the investigators aim to compare platelet inhibition achieved in patients loaded with ticagrelor followed by cangrelor (bolus plus infusion) vs ticagrelor alone loaded patients.

This will be a prospective, randomized, 3-center, single-blind, investigator-initiated study of parallel design to compare platelet inhibition provided by ticagrelor LD plus cangrelor (bolus and infusion) vs ticagrelor LD alone. Participants will be consecutive P2Y12 inhibitor-naive STEMI patients with pain onset<12 hours admitted for primary PCI will be considered.

Participants in both arms will receive ticagrelor 180 mg LD as early as possible (e.g. in the spoke hospital in case of transfer or at the emergency department in cases of hub hospital presentation), as per local practice. The exact time of ticagrelor administration will be recorded. Randomization followed by immediate initiation of cangrelor administration will be performed after angiography and immediately prior to PCI. Patients will be randomized (Hour 0) in a 1:1 ratio by an independent investigator to cangrelor 30 mcg/kg bolus + 4 mcg/kg/min for 2 hours, or no IV antiplatelet .

Other treatment will be as per local standard of care in all participants. Investigators who will perform platelet function testing will be blind to the actual treatment assignment, whereas an independent investigator will monitor bleeding and adverse event data.

Platelet reactivity will be measured at randomization (Hour 0) and at 15 min, 1, 2 and 4 hours post randomization. Platelet function testing will be performed with the VerifyNow (Accumetrics Inc, San Diego, CA) point-of-care P2Y12 function assay within 30 min from blood sample collection. Platelet reactivity results will be reported in P2Y12 reaction units (PRU) and % inhibition. The % inhibition is calculated as: ([BASE-PRU]/BASE)×100. High platelet reactivity (HPR) will be defined as ≥208 PRU.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive P2Y12 inhibitor-naive STEMI patients with pain onset<12 hours admitted for primary PCI.

Exclusion Criteria:

* a history of stroke/transient ischemic attack
* bleeding diathesis
* chronic oral anticoagulation treatment
* contraindications to anti platelet therapy
* PCI or coronary artery bypass grafting <3 months
* platelet count <100 000/μL
* hematocrit <30%
* creatinine clearance <30 mL/min
* severe hepatic dysfunction
* use of strong CYP3A inhibitors or inducers
* increased risk of bradycardia
* severe chronic obstructive pulmonary disease
* periprocedural IIb/IIIa inhibitor administration.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-12-26 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity between the 2 arms | 15 min
  Platelet reactivity in P2Y12 reaction units by VerifyNow assay

SECONDARY OUTCOMES:
Platelet reactivity between the 2 arms | 1 hour
  Platelet reactivity in P2Y12 reaction units by VerifyNow assay
Platelet reactivity between the 2 arms | 2 hours
  Platelet reactivity in P2Y12 reaction units by VerifyNow assay
Platelet reactivity between the 2 arms | 4 hours
  Platelet reactivity in P2Y12 reaction units by VerifyNow assay
High on treatment platelet reactivity rate | 15 min
  High on treatment platelet reactivity rate
High on treatment platelet reactivity rate | 1 hour
  High on treatment platelet reactivity rate
High on treatment platelet reactivity rate | 2 hours
  High on treatment platelet reactivity rate
High on treatment platelet reactivity rate | 4 hours
  High on treatment platelet reactivity rate

OTHER OUTCOMES:
major adverse cardiac events (death, myocardial infarction, stroke, ischemia driven revascularization) | 30 days
Bleeding events (BARC classification) | 30 days
Other adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Alexopoulos, MD, Principal Investigator — Attikon Hospital
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No